CLINICAL TRIAL: NCT04130022
Title: Ultrasound Assessment of Gastric Volume After Drinking Premedication: A Prospective Descriptive Study
Brief Title: Premedication Gastric Ultrasound
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Kevin Spellman (Other)
Responsible Party: Sponsor-Investigator, Kevin Spellman, Anesthesiologist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000586
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fasted Children (Other)
  Interventions: Device: Point-of-Care Ultrasound

INTERVENTIONS:
Device: Point-of-Care Ultrasound — Portable ultrasonography done at the bedside.

SUMMARY:
The primary objective of this study is to assess gastric volume in fasted children using ultrasound before and after drinking premedication. The hypothesis is that the qualitative and quantitative assessment by gastric ultrasound in the stomach before and after drinking premedication will be the same as premedication has a small volume.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 patients aged 0-18 years of scheduled for elective surgery under general anesthesia.

Exclusion Criteria:

* Patients who are not adhere to institutional fasting guidelines.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of Qualitative and Quantitative Gastric Assessment After Premedication | Ultrasound scan performed at baseline (before surgery) to measure gastric volume and 3 minutes after taking premedication to assess change.
  Gastric volume in fasted children before and after drinking premedication. Gastric volume in pediatric patients is estimated by the model: GV= -7.8 + (3.5× RLD CSA) + (0.127) × age (months).

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No